CLINICAL TRIAL: NCT03644589
Title: A Phase II Trial Evaluating Safety and Efficacy of Pembrolizumab and Cisplatin in Patients With Advanced Triple Negative Breast Cancer
Brief Title: Effect of Pembrolizumab and Cisplatin on Metastatic, Locally Recurrent or Inoperable Triple-Negative Breast Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No participants enrolled.
Sponsor: University of Washington (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RG1718047; 9852/MK-3475-315 (Other: FHCRC)
Record Dates: First submitted 2018-08-22; First posted 2018-08-23 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Estrogen Receptor Negative; HER2/Neu Negative; Metastatic Breast Cancer; Progesterone Receptor Negative; Recurrent Breast Carcinoma; Triple Negative Breast Cancer
Keywords: Cisplatin; Pembrolizumab; Keytruda; Triple Negative Breast Cancer; Immune-Checkpoint Inhibitor; Metastatic Breast Cancer; Breast Carcinoma; Recurrent Breast Cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — pembrolizumab; Immunoglobulin G; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (pembrolizumab, cisplatin) (Experimental): Participants receive pembrolizumab and cisplatin once every 3 weeks for a total of 6 doses. Both drugs are given by vein (IV). Participants that are responding to the study treatment will continue to receive pembrolizumab alone beyond 6 cycles for up to 24 months until disease gets worse, having bad side effects, no longer wish to be in the study, or have become pregnant (whichever comes first).
  Participants receive pembrolizumab over 30 minutes and cisplatin on day 1. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. Participants without disease progression after 6 courses may continue on pembrolizumab IV on day 1 every 21 days for up to 24 months (or 35 courses) in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Pembrolizumab; Drug: Cisplatin

INTERVENTIONS:
Biological: Pembrolizumab — 200mg,Given intravenous (IV) infusion, every 21 days
  Other Names: Immunoglobulin G4; Anti-(Human Programmed Cell Death 1); MK-3475
Drug: Cisplatin — 75mg/m2, intravenous (IV) infusion, every 21 days, for 6 cycles Given IV
  Other Names: CDDP

SUMMARY:
This is a Phase II treatment study that is done to evaluate how effective and safe the combination of pembrolizumab and cisplatin work in treating participants with triple-negative breast cancer that had spread to other parts of the body, has come back, or cannot be removed by surgery. Pembrolizumab (investigational drug) is a monoclonal antibody that works by helping your immune system to fight cancer. Cisplatin is a chemotherapy drug that works by interfering with tumor cell division. Studies also suggest that treatment with chemotherapy, like cisplatin, may improve the effectiveness of pembrolizumab. This study will test the effectiveness of pembrolizumab and cisplatin in participants with advanced triple-negative breast cancer.

DETAILED DESCRIPTION:
Participants will receive pembrolizumab intravenously (IV) over 30 minutes and cisplatin once every 3 weeks for a total of 6 doses. Both drugs are given by vein (Intravenous(IV)) on day 1. Participants that are responding to the study treatment will continue to receive pembrolizumab alone for up to 24 months until disease gets worse, having bad side effects, no longer wish to be in the study, or have become pregnant (whichever comes first).

In addition to study drug administration visits, participants will be asked to have physical exams, blood draws every three weeks and tumor evaluation using MRI or CT scans every 9 weeks.

After completion of study treatment, participants are followed up for safety within at 30 days of last dose of study treatment and then every 12 weeks until study completion.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically confirmed diagnosis of metastatic or locally recurrent and inoperable triple negative breast cancer (estrogen receptor [ER] < 10%, progesterone receptor [PR] < 10% and HER2 negative by IHC or fluorescence in situ hybridization [FISH]).
* Be willing and able to provide written informed consent for the trial.
* Have measurable disease based on RECIST 1.1.
* Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on day 1. Participants for whom newly-obtained samples cannot be provided (e.g. inaccessible or participant safety concern) may submit an archived specimen only upon agreement from the principal investigator. * Participants that are screening for second course phase (retreatment period) do not need to comply with the tumor tissue collection eligibility criteria.
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) performance scale. Evaluation of ECOG is to be performed within 10 days prior to the date of treatment initiation.
* Absolute neutrophil count (ANC) >= 1500/uL, performed within 10 days of treatment initiation.
* Platelets >= 100 000/uL, performed within 10 days of treatment initiation.
* Hemoglobin >= 9.0 g/dL or >= 5.6 mmol/L, performed within 10 days of treatment initiation.
* Creatinine =< 1.5 x upper limit of normal (ULN) OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) >= 30 mL/min for participant with creatinine levels > 1.5 x institutional ULN, performed within 10 days of treatment initiation.
* Total bilirubin =< 1.5 x ULN OR direct bilirubin =< ULN for participants with total bilirubin levels > 1.5 x ULN, performed within 10 days of treatment initiation.
* Aspartate aminotransferase (AST) serum glutamic oxaloacetic transaminase ([SGOT]) and alanine aminotransferase (ALT) serum glutamate pyruvate transaminase ([SGPT]) =< 2.5 x ULN (=< 5 x ULN for participants with liver metastases), performed within 10 days of treatment initiation.
* International normalized ratio (INR) OR prothrombin time (PT) =< 1.5 x ULN unless participant is receiving anticoagulant therapy as long as PT or activated partial thromboplastin time (aPTT) is within therapeutic range of intended use of anticoagulants, performed within 10 days of treatment initiation.
* Activated partial thromboplastin time (aPTT) =< 1.5 x ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants, performed within 10 days of treatment initiation.
* Female participants of childbearing potential should have a negative serum pregnancy test performed at the screening visit and a urine pregnancy test performed on cycle 1 day 1 (within 72 hours of receiving the first dose of study medication). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies: * Not a woman of childbearing potential (WOCBP), OR * A WOCBP who agrees to follow the contraceptive guidance during the treatment period and for at least 120 days after the last dose of study treatment. ** Note: abstinence is acceptable if this is the usual lifestyle and preferred contraception for the participant.
* A male participant must agree to use a contraception during the treatment period and for at least 120 days after the last dose of study treatment and refrain from donating sperm during this period. * Note: abstinence is acceptable if this is the usual lifestyle and preferred contraception for the participant.

Exclusion Criteria:

* Has received greater than 3 lines of cytotoxic chemotherapy for metastatic breast cancer.
* Documented disease progression on prior cisplatin therapy.
* Is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment. * Note: participants who have entered the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of study drug.
* Has had a prior monoclonal antibody within 4 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
* Has received prior systemic anti-cancer therapy including investigational agents within 2 weeks prior to first dose of study treatment. * Note: participants must have recovered from all adverse events (AEs) due to previous therapies to =< grade 1 or baseline. Participants with =< grade 2 neuropathy may be eligible. * Note: if participant received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study treatment.
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ) that has undergone potentially curative therapy.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases may participate provided they are radiologically stable, i.e. without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during study screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of study treatment.
* Has severe hypersensitivity (>= grade 3) to pembrolizumab and/or any of its excipients.
* Has received prior radiotherapy within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis. A 1-week washout is permitted for palliative radiation (=< 2 weeks of radiotherapy) to non-CNS disease.
* Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Has an active infection requiring systemic intravenous therapy.
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the participant's participation for the full duration of the trial, or is not in the best interest of the participant to participate, in the opinion of the treating investigator.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
* A WOCBP who has a positive urine pregnancy test within 72 hours prior to first dose of study treatment. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti PD L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137).
* Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies).
* Has a known history of hepatitis B (defined as hepatitis B surface antigen [HBsAg] reactive) or known active hepatitis C virus (defined as hepatitis C virus [HCV] ribonucleic acid (RNA) [qualitative] is detected) infection. * Note: no testing for hepatitis B and hepatitis C is required unless mandated by local health authority.
* Has received a live vaccine within 30 days prior to the first dose of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2021-10-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of combination pembrolizumab and cisplatin in participants with advanced TNBC | Up to 10 years
  Measured by overall response rate (ORR) assessed by RECIST v1.1 criteria.

SECONDARY OUTCOMES:
Safety of pembrolizumab and cisplatin in participants with advanced TNBC | Up to 10 years
  Safety will be assessed by quantifying the toxicities and grades experienced by participants who have received pembrolizumab and cisplatin with summary statistics provided.
Disease Control Rate | Up to 10 years
  Measured by RECIST and irRECIST
Disease control rate (DCR) | Up to 10 years
  Measured by RECIST 1.1 and irRECIST.
Duration of response (DoR) | Up to 10 years
  Measured by RECIST 1.1 and irRECIST
Progression-free survival | Up to 10 years
  Measured by RECIST 1.1 and irRECIST criteria
Overall survival (OS) in participants with advanced TNBC treated with pembrolizumab and cisplatin | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Specht, MD, Principal Investigator — Associate Professor
Locations (1):
- Seattle Cancer Care Alliance, Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No